CLINICAL TRIAL: NCT01559727
Title: Randomized Dose-comparison Study of Prednisone in Patients With Symptomatic Heart Failure
Brief Title: Dose-comparison Study of Prednisone in Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Kun-shen Liu M.D., Professor, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-2011-29
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure
Keywords: heart failure; diuresis; prednisone
MeSH Terms: conditions — Heart Failure | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): The patients with symptomatic heart failure were treated with standard treatment.
- 15 mg prednisone group (Experimental): The patients with symptomatic heart failure are treated with prednisone at dose of 15 mg/day.
  Interventions: Drug: prednisone
- 30 mg prednisone group (Experimental): The patients with symptomatic heart failure are treated with prednisone at dose of 30 mg/day.
  Interventions: Drug: prednisone
- 60 mg prednisone group (Experimental): The patients with symptomatic heart failure are treated with prednisone at dose of 60 mg/day.
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: prednisone — The patients with symptomatic heart failure are treated with prednisone at dose of 15 mg/day.
  Arms: 15 mg prednisone group
Drug: prednisone — The patients with symptomatic heart failure are treated with prednisone at dose of 30 mg/day
  Arms: 30 mg prednisone group
Drug: prednisone — The patients with symptomatic heart failure are treated with prednisone at dose of 60 mg/day
  Arms: 60 mg prednisone group

SUMMARY:
The purpose of this study is to examine the efficacy of three doses of prednisone, a glucocorticoid, in treatment of patients with symptomatic heart failure.

DETAILED DESCRIPTION:
Heart failure is a leading cause of cardiovascular morbidity and mortality in the world. Most patients with acute symptomatic heart failure are admitted with fluid overload. Intravenous loop diuretics are an essential component of current treatment in such patients. Newly emerging evidence showed that glucocorticoids could potentiate natriuretic peptides' action by upregulating the expression natriuretic peptide receptor A (NPR-A) in the kidney, and produce a potent diuresis. Therefore, the investigators designed this nonblinded, randomized dose comparison study to compare the efficacy of prednisone at 15, 30 and 60 mg/day in patients with in symptomatic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized for symptomatic heart failure
* dyspnea at rest or with minimal activity
* NT-proBNP > 1000pg/ml
* LVEF ≤ 40%

Exclusion Criteria:

* any condition (other than CHF) that could limit the use of prednisone;
* acute decompensated heart failure
* active myocarditis
* obstructive or restrictive cardiomyopathy
* cardiac surgery within previous 3 months
* acute coronary syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Daily urinary volumes | 10 days
  Daily urinary volumes will be monitored for 10 days.
Urinary sodium excretion | 10 days
  Daily sodium exretions will be assessed at baseline, day 5 and day 10.

SECONDARY OUTCOMES:
The effect of prednisone on renin angiotensin aldosterone system. | 10 days
  The effect of prednisone on patients' renin angiotensin aldosterone system, such as renin activity, plasma Ang I, plasma Ang II, and plasma aldosterone will be will be assessed on baseline, day 5 and day 10.

CONTACTS AND LOCATIONS:
Overall Officials: Kunshen Liu, MD, Principal Investigator — The First Hospital of Hebei Medical University
Locations (2):
- China (2):
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang

REFERENCES:
- [Derived] Liu C, Zhao Q, Zhen Y, Zhai J, Liu G, Zheng M, Ma G, Wang L, Tian L, Ji L, Li L, Duan L, Liu K. Effect of Corticosteroid on Renal Water and Sodium Excretion in Symptomatic Heart Failure: Prednisone for Renal Function Improvement Evaluation Study. J Cardiovasc Pharmacol. 2015 Sep;66(3):316-22. doi: 10.1097/FJC.0000000000000282. PMID 25992918